CLINICAL TRIAL: NCT04015492
Title: Single Dose, Open Label, Randomized, Cross-over Study in Participants With Severe Hemophilia A Comparing Pharmacokinetic Parameters of BAY 94-9027 and Adynovi
Brief Title: Study to Compare How the Body Distributes and Excretes the Drugs Jivi (BAY 94-9027) and Adynovi in Patients With Severe Hemophilia A (Bleeding Disorder Resulting From a Lack of Blood Clotting Factor VIII)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 19742; 2018-000507-16 (EudraCT Number)
Record Dates: First submitted 2019-07-09; First posted 2019-07-11 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; BAX 855

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BAY94-9027 / Adynovi (Experimental): Treatment sequence A-B with washout before each treatment
  Interventions: Biological: Damoctocog-alfa-pegol (BAY94-9027, Jivi); Biological: Rurioctocog alfa pegol (Adynovi)
- Adynovi / BAY94-9027 (Experimental): Treatment sequence B-A with washout before each treatment
  Interventions: Biological: Damoctocog-alfa-pegol (BAY94-9027, Jivi); Biological: Rurioctocog alfa pegol (Adynovi)

INTERVENTIONS:
Biological: Damoctocog-alfa-pegol (BAY94-9027, Jivi) — Single dose, 50 IU/kg BAY94-9027 (IU: international Units)
Biological: Rurioctocog alfa pegol (Adynovi) — Single dose, 50 IU/kg Adynovi

SUMMARY:
This study is being conducted to compare how the body distributes and excretes the drugs Jivi (BAY 94-9027) and Adynovi. Jivi is a recently approved blood clotting Factor VIII (FVIII) medication for the treatment of hemophilia A (bleeding disorder resulting from a lack of FVIII). Both drugs are FVIII products which have been manufactured via recombinant technology and have an extended half-live, i.e. they will stay longer in the body than other FVIII products. Therefore these products act longer in the body which reduces the frequency of drug injections. To compare the two drugs, a cross-over design was chosen, i.e. each patient will receive both products one after another.

Patients participating in this study will receive one dose of Jivi and one dose of Adynovi. Both drugs are injected into a vein. Observation will last for about 10 weeks, and blood samples will be taken from the participants to measure the blood levels of FVIII. Generic name of Jivi is Damoctocog-alfa-pegol, generic name of Adynovi is Rurioctocog alfa pegol.

ELIGIBILITY:
Inclusion Criteria:

* Participants with severe hemophilia A (baseline FVIII activity FVIII:C <1%), determined by measurement at the time of screening (following a washout period of at least 72 h after their last FVIII treatment for standard half-life FVIII products or of 120 h for extended half-life FVIII products) or from reliable prior documentation (e.g. measurement in other clinical studies, result from approved clinical laboratory or diagnostic genetic testing).
* ≥150 exposure days with FVIII concentrate(s) (plasma-derived or recombinant) as supported by medical records.
* Body mass index (BMI) within the range 18 kg/m2 to 29.9 kg/m2 (inclusive).

Exclusion Criteria:

* Inability to stop FVIII treatment to complete a minimum of 72 h washout for standard half-life FVIII product or 120 h washout for extended half-life FVIII product
* Evidence of current or past inhibitor antibody
* History of any congenital or acquired coagulation disorders other than hemophilia A
* Platelet count <75,000/mm3
* Human immunodeficiency virus (HIV) infection with a cluster of differentiation 4 (CD4+) lymphocyte count of <200/mm3
* Abnormal renal function (serum creatinine >2x the upper limit of the normal range [ULN])
* Active liver disease verified by medical history or persistently elevated alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >5x ULN or severe liver disease as evidenced by, but not limited to any of the following: International Normalized Ratio >1.4, hypoalbuminemia, portal vein hypertension including presence of otherwise unexplained splenomegaly and history of esophageal varices
* Requirement of any pre-medication to tolerate FVIII treatment (e.g. anti-histamines)
* Prior treatment with immunomodulatory agents or chemotherapy within the last 3 months prior to study entry or requirement of treatment during the study. The following drugs are allowed: α interferon, PEG interferon, highly active anti-retroviral therapy for HIV, and/or a total of two courses of pulse treatment with steroid for a maximum of 7 days at 1 mg/kg or less

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2020-01-29 (Actual)

PRIMARY OUTCOMES:
Area under the concentration versus time curve from time 0 to the last data point (AUC(0-tlast)) for BAY 94-9027 | Pre-dose to 120 hours after the end of the infusion
Area under the concentration versus time curve from time 0 to the last data point (AUC(0-tlast)) for Adynovi | Pre-dose to 120 hours after the end of the infusion

CONTACTS AND LOCATIONS:
Locations (1):
- SHATHD Spec. Hospi. for Active Treatm. of Haematol. Dis. EAD, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Solms A, Shah A, Berntorp E, Tiede A, Iorio A, Linardi C, Ahsman M, Mancuso ME, Zhivkov T, Lissitchkov T. Direct comparison of two extended half-life PEGylated recombinant FVIII products: a randomized, crossover pharmacokinetic study in patients with severe hemophilia A. Ann Hematol. 2020 Nov;99(11):2689-2698. doi: 10.1007/s00277-020-04280-3. Epub 2020 Sep 24. PMID 32974838
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/